CLINICAL TRIAL: NCT00384943
Title: Decreasing Health Care Utilization With Alternative Approaches for the Treatment of Depression: A Randomized Trial of Exercise for Postpartum Depression
Brief Title: Study of Home-Based Exercise to Alleviate Postpartum Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FRSQ 024018
Record Dates: First submitted 2006-10-04; First posted 2006-10-06 (Estimated); Last update posted 2006-10-06 (Estimated); Status verified 2006-10

CONDITIONS: Postpartum Depression
Keywords: postpartum depression; exercise
MeSH Terms: conditions — Depression, Postpartum; Motor Activity

INTERVENTIONS:
Behavioral: Moderate-intensity Exercise

SUMMARY:
The purpose of this study is to evaluate the effectiveness of an aerobic home-based exercise program for the treatment of postpartum depression.

DETAILED DESCRIPTION:
Postpartum depression occurs in 10-16% of women, with depressive symptoms lasting up to one year post delivery. Women affected by depression in the postpartum have been shown to be at higher risk for developing a recurrent depressive disorder. While the direct and indirect costs associated with postpartum depression are unknown, those associated with depression have been found to exceed 43 billion dollars in the United States alone. Moreover, maternal depression can negatively impact the mother-infant relationship and infant development. Despite the high prevalence of postpartum depression, the condition often goes undiagnosed and untreated by primary care providers. Alternative non-medical interventions for treating postpartum depression have not been widely investigated, leaving women and health care providers with few evidence-based options for treatment. If this exercise program is shown to be effective, then this intervention can be an alternate treatment option for alleviating depressed mood for women in the postpartum period. This nonpharmacological approach may be particularly attractive as many women are reluctant to take medication in the postpartum.

ELIGIBILITY:
Inclusion Criteria:

* women 4 to 38 weeks following childbirth
* score of 10 or more on the Edinburgh Postpartum Depression Scale
* understand English or French
* no current alcohol or substance abuse,
* not currently participating in regular moderate or high intensity exercise (30 minutes, at least 3 times per week)

Exclusion Criteria:

* obstetrical or concomitant diseases which would have precluded participation in an exercise program.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2001-11; Study Completion 2004-11

PRIMARY OUTCOMES:
Change in depressed mood scores immediately following the 3 month intervention and at 3 and 6 months post-treatment,
as measured by the Edinburgh Postnatal Depression Scale and the Hamilton Rating Scale for Depression.

SECONDARY OUTCOMES:
Changes in fatigue levels (measured by the multidimensional fatigue inventory), sleep patterns, anxiety and health status.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Da Costa, PhD, Principal Investigator — McGill University
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada